CLINICAL TRIAL: NCT07121881
Title: Clinical And Radiographic Evaluation of Mandibular Implant Assisted Overdenture Between Bar Attachment and Bar With OT Equator Attachment: Randomized Controlled Trial
Brief Title: Mandibular Implant Overdenture With Bar vs OT Equator: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hala Abdel salam Selim (Other)
Responsible Party: Sponsor-Investigator, Hala Abdel salam Selim, PhD Candidate, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS-OTBarRCT2024
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-05

CONDITIONS: Edentulous Mandible; Implant-Supported Overdentures
Keywords: OT Equator attachment; Denture retention; Crestal bone loss; Patient satisfaction; Bar attachment; cap wear
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial: Group 1 receives bar attachment only; Group 2 receives bar with OT Equator attachment.
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor (statistician) is blinded to the group allocation. Due to the nature of the interventions, participants and investigators cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bar Attachment Only (Active Comparator): Participants in this group will receive a mandibular implant-assisted overdenture supported by a milled bar attachment only. Three implants will be placed in the anterior mandible (midline and canine regions), and a bar attachment will be fabricated without any additional retentive elements.
  Interventions: Device: Bar Attachment
- Bar with OT Equator Attachment (Experimental): Participants in this group will receive a mandibular implant-assisted overdenture supported by a milled bar with OT Equator attachments. Three implants will be placed in the anterior mandible (midline and canine regions). Two OT Equator attachments will be incorporated into the bar to enhance retention and stress distribution.
  Interventions: Device: Bar with OT Equator Attachment

INTERVENTIONS:
Device: Bar Attachment — A bar attachment supported by three mandibular implants (placed in the midline and canine regions) is used to retain a mandibular overdenture. The bar provides rigid splinting across the implants and allows retention using friction or clips, without additional attachment components. This serves as the control group.
  Arms: Bar Attachment Only
Device: Bar with OT Equator Attachment — A bar attachment supported by three mandibular implants is combined with two OT Equator attachments to enhance denture retention and allow slight vertical and rotational resilience. The OT Equator system includes metal housings and retentive nylon caps, intended to reduce cap wear and improve patient comfort. This is the experimental arm.
  Arms: Bar with OT Equator Attachment

SUMMARY:
This clinical study will evaluate two types of attachment systems used to support lower dentures in patients who have lost all their lower teeth. All participants will receive dental implants in the lower jaw, and a complete denture that attaches to these implants for better stability and comfort.

The study compares two options:

A traditional bar attachment

A bar with additional OT Equator attachments, which are designed to improve denture retention and reduce wear

Each participant will receive three implants in the lower jaw, and either a bar attachment alone or a bar with OT Equator attachments will be placed. The goal is to find out which method provides better retention of the denture, causes less bone loss around the implants, has less wear on the attachment parts, and leads to higher patient satisfaction.

Participants will be followed over several months. Their denture retention will be tested using a digital force meter, bone levels will be measured through radiographs, cap wear will be examined using an electron microscope, and satisfaction will be recorded using a questionnaire.

This study is being conducted at Cairo University and is self-funded by the primary investigator. Participation is voluntary and does not involve any financial cost to participants.

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to compare the clinical and radiographic outcomes of mandibular implant-supported overdentures using two different attachment systems: bar attachment alone (control group) versus bar with OT Equator attachments (intervention group).

A total of 22 completely edentulous participants will be randomly assigned to either group. Each participant will receive three dental implants placed in the anterior mandible. After healing, bar attachments will be fabricated and delivered. In the intervention group, OT Equator attachments will be added to the bar to enhance retention and flexibility. All participants will receive complete upper and lower dentures.

The study's primary outcome is denture retention, measured using a digital force gauge. Secondary outcomes include crestal bone loss (assessed radiographically), cap wear (measured via electron microscopy), and patient satisfaction (evaluated with a Visual Analog Scale questionnaire).

This study will help inform clinical decisions regarding attachment systems for mandibular overdentures and may provide evidence for improved long-term function and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous healthy patients.
* Age between 35 and 65 years.
* Sufficient bone in the anterior and premolar-molar regions (≥11 mm).
* Adequate inter-arch space (12-14 mm).

Exclusion Criteria:

* Severe maxillomandibular skeletal discrepancy.
* Presence of parafunctional habits such as clenching or bruxism.
* Temporomandibular joint disorders.
* Smokers.
* History of drug abuse.
* History of head and neck radiation.
* Systemic disorders that could prevent surgery or affect bone quality (e.g., uncontrolled diabetes, osteoporosis).

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Retention of Mandibular Overdenture | At baseline (T0) and 6 months post-insertion (T6)
  Retention will be measured using a digital force gauge. A standardized technique will be used to measure the force required to dislodge the mandibular overdenture by pulling upward from a geometric center marked on the denture.

SECONDARY OUTCOMES:
Crestal Bone Loss Around Implants | At baseline (T0) and 6 months post-insertion (T6)
  Bone level changes will be assessed radiographically using the long cone parallel technique. Crestal bone height will be measured on standardized radiographs at two time points and recorded in millimeters.
Cap Wear of Attachment System | At baseline (T0) and 6 months post-insertion (T6)
  Cap wear will be evaluated by measuring physical changes in the nylon caps of the attachments using an electron microscope. Measurements will be taken in millimeters to assess material degradation.
Patient Satisfaction | At 6 months post-insertion (T6)
  Patients will complete a Visual Analog Scale (VAS) questionnaire assessing overall satisfaction, comfort, speech, chewing ability, aesthetics, and ease of cleaning with the overdenture.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Abo EL-Fotouh, Professor, Study Chair — Faculty of Oral and Dental Medicine, Cairo University; Noha Ali, asso. Professor, Study Director — Faculty of Oral and Dental Medicine, Cairo University; Ahmed Hamed, Lecturer, Study Director — Faculty of Oral and Dental Medicine, Cairo University
Locations (1):
- Faculty of Oral and Dental Medicine, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant confidentiality and because no formal mechanisms are in place for data sharing beyond the study team. Data will remain securely stored at Cairo University and accessible only to the authorized research team.